CLINICAL TRIAL: NCT00812435
Title: Eptifibatide and ST Segment Resolution Following Primary PCI
Acronym: ESTEEM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESTEEM
Record Dates: First submitted 2008-02-17; First posted 2008-12-22 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Myocardial Infarction
Keywords: STEMI; Patients; male or female; greater than 18 years of age; presenting with ST elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eptifibatide (Experimental): PCI with administration of eptifibatide
  Interventions: Drug: eptifibitide

INTERVENTIONS:
Drug: eptifibitide — Patients will be randomized to eptifibatide or no eptifibatide. If randomized to eptifibatide: 180 mcg/kg Bolus; 2 mcg/kg/min infusion immediately prior to primary PCI or at the time of PCI and for 18 - 24 hours following the PCI Second 180 mcg/kg Bolus 10 min after the first
  Other Names: Integrilin

SUMMARY:
This is a prospective, open label, randomized trial of 100 patients who present to the cardiac catheterization laboratory with an ST Elevation Myocardial Infarction for primary PCI. Patients may receive up-front unfractionated heparin or low molecular weight heparin, but not glycoprotein IIb/IIIa inhibitors or thrombolytics. Patients will be consented prior to the diagnostic catheterization and will be randomized once the patient is deemed amenable to PCI to receive eptifibatide or no eptifibatide just prior to or at the time of primary angioplasty. Patients will be randomized in a 1:1 fashion. All patients will be assessed for the primary endpoint of ST resolution at 60 minutes post PCI and followed throughout the duration of the hospitalization and up to 30 days for secondary endpoint evaluation.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness and safety of adjunctive eptifibatide during primary PCI in patients presenting to the catheterization laboratory within 12 hours of symptom onset. The primary objective of this randomized clinical trial is to examine the safety and effectiveness of the addition of eptifibatide therapy immediately prior to or at the time of PCI in patients presenting with a STEMI for primary PCI who have not received up-front glycoprotein IIb/IIIa inhibitor therapy. The secondary objective of this clinical trial is to assess effectiveness of adjunct eptifibatide therapy with respect to the following endpoints:

* Complete ST resolution (defined above) at 90 and 180 minutes post primary PCI
* TIMI flow at the end of the PCI (as reported by the investigator at the end of the procedure)
* MACE evaluation at discharge and 30 days post PCI (MACE defined as: death, reinfarction, and need for urgent ischemia-driven target vessel revascularization)
* Stent thrombosis at discharge and 30 days
* Major Bleed (Major Bleed defined as: TIMI Major Bleeding)
* Minor Bleed (Minor Bleed defined as: TIMI Minor Bleeding)
* ST segment resolution at 60, 90 and 180 minutes based on the additional measure in the Schroder's Index:
* Partial resolution defined as 30-70% ST-segment resolution, and
* No resolution defined as <30% ST-segment resolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Patients with acute myocardial infarction whose symptom onset is within 12 hours of presentation
* ST-segment elevation 1 mm in 2 contiguous limb leads or 2 mm in 2 contiguous precordial leads
* Patients eligible for PCI
* Target lesion(s) in a native vessel
* Target lesion stenosis >50% by angiography (visual estimate)
* Patients who are amenable to participating in study procedures and follow-up
* Patient or legal guardian has been informed and agrees to provide approved written informed consent and data privacy authorization

Exclusion Criteria:

* Patients with cardiogenic shock (SBP<80 mmHg for >30 minutes or requiring pressors or IABP due to hypotension)
* Patients with cardiac arrest at any point prior to intervention (within the preceeding 24 hours)
* Patients on chronic warfarin (Coumadin) therapy
* Patients with known bleeding diathesis or active bleeding at the time of presentation to the catheterization laboratory
* Patients with known bleeding diathesis or active bleeding within prior 3 months
* Patients who receive thrombolytic therapy or glycoprotein IIb/IIIa inhibitors prior to PCI (within the preceding 8 hours)
* Patients with a platelet count <100,000 cells/mm3 within the preceeding 7 days
* Patients with known allergies to aspirin, clopidogrel bisulfate (Plavix), heparin, bivalirudin, glycoprotein IIb/IIIa inhibitors or intravenous contrast dye that cannot be medically managed
* Patients with major surgery within the past 6 months or scheduled surgery within 6 weeks
* Patients with significant unprotected left main disease (stenosis >60%) or with multivessel coronary disease that will require emergent coronary artery bypass surgery
* Patients with TIA or CVA within the past 30 days or any history of hemorrhagic stroke
* Patients who have undergone PCI within the preceding 30 days prior to enrollment
* Patients with known impaired renal function
* Patient is know to be pregnant or lactating
* Patients with active participation in another device or drug study
* Patients with comorbidities conferring a life expectancy of less than a year
* Patients with left bundle branch block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2010-07 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be complete ST resolution 60 minutes following primary PCI where complete ST resolution is defined as ≥70% ST resolution compared to the qualifying ECG. | In patient hopsitalization

SECONDARY OUTCOMES:
Complete ST resolution (defined above) at 90 and 180 minutes following primary PCI; TIMI flow at the end of the PCI; and MACE evaluation at discharge and 30 days post PCI | In-patient hospitalization and 30 days post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States